CLINICAL TRIAL: NCT00485953
Title: The Effect of Bisphosphonate on Bone Mass and Bone Turnover in Elderly, Postmenopausal Women With Breast Cancer Following Initiation of Aromatase Inhibitor Therapy
Brief Title: Effect of Bisphosphonate on Bone Loss in Postmenopausal Women With Breast Cancer Initiating Aromatase Inhibitor Therapy
Acronym: REBBeCA II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Susan L. Greenspan (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Susan L. Greenspan, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO06080002 (REBBeCA II)
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Bone Loss; Osteoporosis; Breast Cancer
Keywords: Osteoporosis; breast cancer; aromatase inhibitors; bone loss; bone mineral density
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Breast Neoplasms | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Medication Group (Experimental): risedronate 35 mg weekly
  Interventions: Drug: risedronate
- Placebo Group (No Intervention): Placebo

INTERVENTIONS:
Drug: risedronate — risedronate 35 mg per week
  Other Names: Actonel
  Arms: Active Medication Group

SUMMARY:
Elderly, postmenopausal women with breast cancer on aromatase inhibitors are at increased risk of developing bone loss and osteoporosis. We postulate that in elderly, osteopenic postmenopausal women who are on aromatase inhibitor therapy, bisphosphonate therapy will (1) prevent bone loss at clinically relevant sites, such as the spine and hip and (2) decrease bone turnover.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled, randomized clinical trial will test the hypothesis that risedronate 35 mg once weekly, a potent antiresorptive agent, will prevent bone loss or improve bone mass and decrease bone turnover in elderly, osteopenic, postmenopausal women (ages 55 and older) with breast cancer on aromatase inhibitor therapy. 110 subjects will be randomized to receive either oral risedronate 35 mg once weekly or placebo for two years. Our primary outcome variable will be change in PA spine bone mineral density (BMD). Secondary endpoints will be BMD at the total hip, femoral neck, trochanter, lateral spine, forearm, and total body, and markers of bone turnover. We will also assess if the improvements in BMD are greater at sites of trabecular bone (spine) versus cortical bone (wrist). BMD will be measured at six month intervals. Biochemical markers of bone turnover will be measured at baseline, 6 months, 12 months, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* elderly postmenopausal women (ages 55 and older)
* osteopenic (DXA T-score -1.0 to -2.5 SD). However, after full counseling about the risks, benefits, and options regarding therapy for osteoporosis and discussion with her PCP, an osteoporotic woman may enroll in the study.
* with breast cancer on aromatase inhibitor therapy
* with no evidence of distant metastatic disease or osteoporosis (by BMD or clinical history)
* type of surgical procedure or addition of radiation therapy prior to this aromatase inhibitor therapy will not exclude patients
* Participants must provide voluntary, written informed consent to participate in the study, which includes understanding of the procedures, medications, and risks and benefits

Exclusion Criteria:

* Women with stage 4 breast cancer (presence of distant metastases)
* Women with normal bone density by DXA (T-score > -1.0 SD)bone density by DXA, except in the instance of a fragility fracture.
* Women with history of any illness known to affect bone and mineral metabolism, such as renal failure (estimated GFR <30), hepatic failure, malignancy (excluding breast cancer, treated superficial basal and squamous cell carcinoma and malignancies where the diagnosis itself or its treatment would not adversely affect bone metabolism), untreated primary hyperparathyroidism, and malabsorption.
* Women being treated with oral glucocorticoid therapy >3 months for suppression therapy, and certain anti-seizure medications which may adversely affect bone metabolism (phenobarbital, phenytoin, carbamazepine).
* Those with untreated active peptic ulcer disease
* Those with osteoporosis by BMD (T-score -2.5 SD at the spine or total hip) or a history of fragility fracture as an adult. However, as discussed above, osteoporotic women may elect to enroll in the study.
* Women treated with oral bisphosphonates or calcitonin for 3 months within the last year (3 month washout period)
* Men and children will be excluded because they do not get postmenopausal osteoporosis following treatment with an aromatase inhibitor
* Women with very poor dental hygiene (as assessed by the baseline dental exam) in need of dental extraction during the study
* Use of fluoride for more than 1 month ever (except for dental treatment)
* Less than 2 evaluable vertebrae
* Distant metastatic disease

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2007-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L. Greenspan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: Received placebo medication once per week
Period: Overall Study
Arm/Group | Active Medication Group | Placebo Group
Started | 55 | 54
Completed | 48 | 47
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Active Medicine Group: risedronate 35 mg weekly
- Total: Total of all reporting groups
Arm/Group | Active Medicine Group | Placebo Group | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 34 | 66
  >=65 years | 23 | 20 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 54 | 109
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 47 | 53 | 100
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 55 | 53 | 108
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 54 | 109

OUTCOME MEASURES:

1. Primary Outcome: BMD of Spine by DXA
Description: BMD is the bone mineral density of the lumbar spine measured using the dual-energy x-ray absorptometry (DXA) scan.
Time Frame: at 24 months
Measure: Mean (Standard Error); unit: percentage change
Groups:
- Placebo Group: Received placebo medication once weekly
Arm/Group | Active Medicine Group | Placebo Group
Number analyzed (Participants) | 55 | 54
percentage change | 2.269 (0.583) | -1.735 (0.611)

2. Secondary Outcome: BMD by DXA at the Femoral Neck and Total Hip
Description: BMD is the bone mineral density of the femoral neck and total hip measured using the dual-energy x-ray absorptiometry (DXA) scan.
Time Frame: at 24 months
Measure: Mean (Standard Error); unit: percentage change
Groups:
- Placebo Group: Placebo medication once weekly
Arm/Group | Active Medication Group | Placebo Group
Number analyzed (Participants) | 47 | 44
percentage change
  Total Hip BMD | 0.558 (0.370) | -2.748 (0.487)
  Femoral Neck BMD | 0.408 (0.607) | -2.137 (0.628)

3. Secondary Outcome: Markers of Bone Resorption and Bone Formation
Time Frame: at 24 months
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Active Medicine Group | Placebo Group
Number analyzed (Participants) | 48 | 47
percentage change
  CTX | -14.906 (10.317) | -4.077 (8.179)
  P1NP | -46.863 (3.025) | -1.630 (5.732)

ADVERSE EVENTS:
Groups:
- Placebo Group: Receive placebo medication once per week
Arm/Group | Active Medicine Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 10/55 | 16/54
Other Adverse Events (participants affected / at risk) | 52/55 | 50/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Medicine Group (N=55) | Placebo Group (N=54)
Breast related events (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Gastrointestinal Events (Gastrointestinal disorders) | 0 (0) | 1 (1)
Respiratory related events (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cardiovascular related events (Cardiac disorders) | 5 (5) | 2 (2)
Musculoskeletal related events (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Infection related events (Infections and infestations) | 2 (2) | 3 (3)
Urogenital related events (Renal and urinary disorders) | 0 (0) | 1 (1)
Other cancers (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Other events (General disorders) | 0 (0) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Medicine Group (N=55) | Placebo Group (N=54)
Breast related events (Reproductive system and breast disorders) | 4 (4) | 3 (3)
Gastrointestinal related events (Gastrointestinal disorders) | 4 (4) | 12 (12)
Respiratory related events (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (10)
Cardiovascular related events (Cardiac disorders) | 4 (4) | 10 (10)
Musculoskeletal related events (Musculoskeletal and connective tissue disorders) | 27 (27) | 32 (32)
Infection related events (Infections and infestations) | 13 (13) | 14 (14)
Endocrine related events (Endocrine disorders) | 2 (2) | 4 (4)
Urogenital related events (Renal and urinary disorders) | 3 (3) | 6 (6)
Other cancers (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Other events (General disorders) | 26 (26) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes